CLINICAL TRIAL: NCT03486314
Title: A Phase 1 Study to Evaluate the Effects of Rifampin on Pharmacokinetics of Pevonedistat in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Effects of Rifampin on Pharmacokinetics (PK) of Pevonedistat in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Pevonedistat-1015; U1111-1202-2144 (Other: WHO)
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Results first posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-02

CONDITIONS: Advanced Solid Neoplasm
Keywords: Drug therapy
MeSH Terms: interventions — pevonedistat; Rifampin; Docetaxel; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg (Experimental): Pevonedistat 50 milligram per square meter (mg/m^2), intravenous infusion, once on Day 1 and 10 along with rifampin 600 milligram (mg), capsule, orally, once daily from Day 3 up to Day 11 in Part A. After completion of Part A, participants had opportunity to continue into optional Part B.
  Interventions: Drug: Pevonedistat; Drug: Rifampin
- Part B: Pevonedistat (Experimental): Pevonedistat 25 mg/m^2 intravenously in combination with docetaxel 75 mg/m^2 or at 20 mg/m^2 in combination with carboplatin +paclitaxel 175 mg/m^2; pevonedistat was given in combination on Day 1 and as a single agent on Days 3 and 5 of each 21-day cycle. Participants were treated for up to 12 cycles or symptomatic deterioration or PD, treatment was discontinued for another reason, or until the study is stopped in Part B. The choice of combination partner (docetaxel or carboplatin + paclitaxel) was based on investigator discretion. If the sponsor and investigator determine that a participant would derive clinical benefit from continued treatment, the participant may remain on the current combination therapy or receive pevonedistat as a single agent beyond 12 cycles.
  Interventions: Drug: Pevonedistat; Drug: Docetaxel; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pevonedistat — Pevonedistat intravenous infusion.
  Other Names: MLN4924, TAK-924
Drug: Rifampin — Rifampin capsules.
  Arms: Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg
Drug: Docetaxel — Docetaxel intravenous infusion.
  Arms: Part B: Pevonedistat
Drug: Carboplatin — Carboplatin intravenous infusion.
  Arms: Part B: Pevonedistat
Drug: Paclitaxel — Paclitaxel intravenous infusion.
  Arms: Part B: Pevonedistat

SUMMARY:
The purpose of this study is to assess the effect of multiple-dose administration of rifampin on the single dose PK of pevonedistat in adult participants with advanced solid tumors.

DETAILED DESCRIPTION:
The study will enroll approximately 20 participants. The study will be conducted in two Parts: Part A and optional Part B. Part A will have a drug-drug interaction (DDI) assessment. In Part A, participants will be assigned to:

• Pevonedistat 50 mg/m^2 + Rifampin

Eligible participants from Part A will continue treatment in optional Part B with pevonedistat in combination with SoC chemotherapy, docetaxel or carboplatin plus paclitaxel. The investigator will decide which SoC combination partner a participant will receive.

* Pevonedistat 25 mg/m^2 + Docetaxel
* Pevonedistat 20 mg/m^2 + Carboplatin + Paclitaxel

This multi-center trial will be conducted in the United States. The overall time to participate in this study is 18 months. Participants will make a final visit to the clinic 30 days after receiving their last dose of study drug or before the start of subsequent therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants who have a histologically or cytologically confirmed metastatic or locally advanced solid tumor that is appropriate for treatment with either docetaxel or carboplatin + paclitaxel in Part B of this study, or have progressed despite standard therapy, or for whom conventional therapy is not considered effective.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
3. Expected survival of at least 3 months from the date of enrollment in the study.
4. Recovered (that is, less than or equal to (<=) Grade 1 toxicity) from the effects of prior antineoplastic therapy.
5. Adequate organ functions (kidney, liver, cardiac, bone marrow).
6. Suitable venous access for the study-required blood sampling (including PK sampling).

Exclusion Criteria:

1. Prior treatment with radiation therapy involving greater than or equal to (>=) 25% of the hematopoietically active bone marrow.
2. Life-threatening illness or serious (acute or chronic) medical or psychiatric illness unrelated to cancer.
3. Active, uncontrolled infection or severe infectious disease.
4. Known human immunodeficiency virus (HIV) seropositive or known hepatitis B or hepatitis C infection.
5. With significant heart or pulmonary disease.
6. Requiring chronic treatment with breast cancer resistance protein (BCRP) inhibitors.

Criteria for Continuation into Optional Part B:

To be eligible for Part B, participants must have completed Part A and be reassessed to determine if they meet the continuation criteria for Part B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Greenville Health System - Institute for Translational Oncology Research, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Zhou X, Vaishampayan U, Mahalingam D, Harvey RD, Chung KY, Sedarati F, Dong C, Faller DV, Venkatakrishnan K, Gupta N. Phase 1 study to evaluate the effects of rifampin on pharmacokinetics of pevonedistat, a NEDD8-activating enzyme inhibitor in patients with advanced solid tumors. Invest New Drugs. 2022 Oct;40(5):1042-1050. doi: 10.1007/s10637-022-01286-8. Epub 2022 Aug 6. PMID 35932388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 13 August 2018 to 28 February 2021.
Pre-assignment Details: Participants with histologically or cytologically confirmed metastatic or locally advanced solid tumor were enrolled in this 2-part study to receive intravenous infusion of pevonedistat along with rifampin capsule in Part A and pevonedistat in combination with chemotherapy agents in Part B (optional part). After completion of Part A, participants had an opportunity to continue into optional Part B.
Groups:
- Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg: Pevonedistat 50 milligram per square meter (mg/m^2), infusion, intravenously, once on Days 1 and 10, and then rifampin 600 milligram (mg), capsule, orally, once daily from Day 3 up to Day 11 in Part A. Pevonedistat was not administered from Day 2 through Day 9.
- Part B: Pevonedistat 25 mg/m^2 + Docetaxel 75 mg/m^2: Pevonedistat 25 mg/m^2, infusion, intravenously in combination with docetaxel 75 mg/m^2, infusion, intravenously on Day 1 of 21-day cycle, followed by pevonedistat 25 mg/m^2, infusion, intravenously alone once on Days 3 and 5 in each 21-day cycle for up to 17 cycles or symptomatic deterioration or disease progression, treatment discontinuation for another reason, or until the study was stopped in Part B. Participants who completed Part A and provided consent for Part B continued treatment in Part B.
- Part B: Pevonedistat 20 mg/m^2 + Carboplatin AUC5+ Paclitaxel 175 mg/m^2: Pevonedistat 20 mg/m^2, infusion, intravenously in combination with carboplatin area under the plasma concentration (AUC) at the dose of 5 milligram* minute per milliliter (mg*min/mL), infusion, intravenously and paclitaxel 175 mg/m^2, infusion, intravenously, once on Day 1 of 21-day cycle, followed by pevonedistat 20 mg/m^2, infusion, intravenously alone once on Days 3 and 5 in each 21-day cycle for up to 17 cycles or symptomatic deterioration or disease progression, treatment was discontinued for another reason, or until the study was stopped in Part B. Pevonedistat was administered after the paclitaxel and carboplatin chemotherapy. Participants who completed Part A and provided consent for Part B continued treatment in Part B.
Period: Part A
Arm/Group | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg | Part B: Pevonedistat 25 mg/m^2 + Docetaxel 75 mg/m^2 | Part B: Pevonedistat 20 mg/m^2 + Carboplatin AUC5+ Paclitaxel 175 mg/m^2
Started | 20 | 0 | 0
Completed | 17 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Symptomatic Deterioration | 2 | 0 | 0
Period: Part B
Arm/Group | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg | Part B: Pevonedistat 25 mg/m^2 + Docetaxel 75 mg/m^2 | Part B: Pevonedistat 20 mg/m^2 + Carboplatin AUC5+ Paclitaxel 175 mg/m^2
Started | 0 | 9 (These are the participants who completed Part A, met eligibility criteria, and provided consent for Part B.) | 8 (These are the participants who completed Part A, met eligibility criteria, and provided consent for Part B.)
Completed | 0 | 9 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set for Part A was defined as all enrolled participants who received at least a single pevonedistat dose during Part A.
Groups:
- Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg: Pevonedistat 50 mg/m^2, infusion, intravenously, once on Days 1 and 10, and then rifampin 600 mg, capsule, orally, once daily from Day 3 up to Day 11 in Part A. Pevonedistat was not administered from Day 2 through Day 9.
Arm/Group | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 171.91 (10.235)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 87.13 (22.667)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meter (m^2)] | 2.03 (0.307)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Ratio of Maximum Observed Plasma Concentration (Cmax) for Pevonedistat Without Rifampin (Day 1) and With Rifampin (Day 10)
Description: The Least square (LS) means ratio of Day 10 over Day 1 were calculated from a mixed-model analysis of variance model.
Time Frame: Days 1 and 10 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The pharmacokinetic (PK) evaluable population was defined as all enrolled participants who a) received the protocol specified single pevonedistat dose in Part A; b) did not receive any excluded medications throughout the completion of Part A; and c) had sufficient concentration-time data to permit reliable estimation of PK parameters. As planned, this outcome measure was only assessed in Part A. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg
Number analyzed (Participants) | 17
ratio | 0.962 [0.792 to 1.168]

2. Primary Outcome: Part A: Ratio of Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for Pevonedistat Without Rifampin (Day 1) and With Rifampin (Day 10)
Description: The LS means ratio of Day 10 over Day 1 were calculated from a mixed-model analysis of variance model.
Time Frame: Days 1 and 10 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The PK-evaluable population was defined as all enrolled participants who a) received the protocol specified single pevonedistat dose in Part A; b) did not receive any excluded medications throughout the completion of Part A; and c) had sufficient concentration-time data to permit reliable estimation of PK parameters. As planned, this outcome measure was only assessed in Part A. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg
Number analyzed (Participants) | 17
ratio | 0.785 [0.684 to 0.901]

3. Primary Outcome: Part A: Ratio of Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC∞) for Pevonedistat Without Rifampin (Day 1) and With Rifampin (Day 10)
Description: The LS means ratio of Day 10 over Day 1 were calculated from a mixed-model analysis of variance model.
Time Frame: Days 1 and 10 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg
Number analyzed (Participants) | 17
ratio | 0.790 [0.692 to 0.902]

4. Secondary Outcome: Part A: Total Clearance After Intravenous Administration (CL) for Pevonedistat Without Rifampin (Day 1) and With Rifampin (Day 10)
Time Frame: Days 1 and 10 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The PK-evaluable population was defined as all enrolled participants who a) received the protocol specified single pevonedistat dose in Part A; b) did not receive any excluded medications throughout the completion of Part A; and c) had sufficient concentration-time data to permit reliable estimation of PK parameters. As planned, this outcome measure was only assessed in Part A. Here number analyzed "n" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg
Number analyzed (Participants) | 20
liter per hour (L/h)
  Pevonedistat without rifampin (Day 1) | 35.22 (10.980)
  Pevonedistat with rifampin (Day 10): number analyzed (Participants) | 17
  Pevonedistat with rifampin (Day 10) | 43.77 (12.604)

5. Secondary Outcome: Part A: Volume of Distribution at Steady State After Intravenous Administration (Vss) for Pevonedistat Without Rifampin (Day 1) and With Rifampin (Day 10)
Time Frame: Days 1 and 10 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg
Number analyzed (Participants) | 20
liter
  Pevonedistat without rifampin (Day 1) | 312.82 (144.495)
  Pevonedistat with rifampin (Day 10): number analyzed (Participants) | 17
  Pevonedistat with rifampin (Day 10) | 296.10 (136.297)

6. Secondary Outcome: Part A: Terminal Disposition Phase Half-life (T1/2z) for Pevonedistat Without Rifampin (Day 1) and With Rifampin (Day 10)
Time Frame: Days 1 and 10 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg
Number analyzed (Participants) | 20
hour
  Pevonedistat without rifampin (Day 1) | 7.442 (1.3846)
  Pevonedistat with rifampin (Day 10): number analyzed (Participants) | 17
  Pevonedistat with rifampin (Day 10) | 5.708 (1.3665)

7. Secondary Outcome: Part B: Number of Participants With Best Overall Response as Per Investigator's Assessment
Description: Best overall response was defined as participants with best response among complete response (CR) or partial response (PR) or stable disease (SD), or progressive disease (PD). It was assessed by investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target and non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR: at least 30 percent (%) decrease in sum of diameter of target lesions, taking as reference baseline sum of diameter. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum of diameter. PD: at least 20% increase in sum of diameter of target lesions, taking as reference, smallest sum on study.
Time Frame: Up to Cycle 17 (end of treatment) (Cycle length =21 days)
Population: The response-evaluable population was defined as all participants who received at least 1 dose of study drug in Part B, had measurable disease as entry criteria for Part B, and had at least 1 postbaseline disease assessment. As planned, this outcome measure was only assessed in Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Pevonedistat 20 mg/m^2 + Carboplatin AUC5 + Paclitaxel 175 mg/m^2: Pevonedistat 20 mg/m^2, infusion, intravenously in combination with carboplatin AUC at the dose of 5 mg*min/mL, infusion, intravenously and paclitaxel 175 mg/m^2, infusion, intravenously, once on Day 1 of 21-day cycle, followed by pevonedistat 20 mg/m^2, infusion, intravenously alone once on Days 3 and 5 in each 21-day cycle for up to 17 cycles or symptomatic deterioration or disease progression, treatment was discontinued for another reason, or until the study was stopped in Part B. Pevonedistat was administered after the paclitaxel and carboplatin chemotherapy. Participants who completed Part A and provided consent for Part B continued treatment in Part B.
Arm/Group | Part B: Pevonedistat 25 mg/m^2 + Docetaxel 75 mg/m^2 | Part B: Pevonedistat 20 mg/m^2 + Carboplatin AUC5 + Paclitaxel 175 mg/m^2
Number analyzed (Participants) | 6 | 7
Participants
  CR | 0 | 0
  PR | 2 | 1
  SD | 2 | 3
  PD | 2 | 3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (From first dose of study drug up to Day 41 [Part A]; From first dose of study drug up to Cycle 17 Day 35 (Cycle length =21 days) [Part B])
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Part B: Pevonedistat 20 mg/m^2 + Carboplatin AUC5+ Paclitaxel 175 mg/m^2: Pevonedistat 20 mg/m^2, infusion, intravenously in combination with carboplatin AUC at the dose of 5 mg*min/mL, infusion, intravenously and paclitaxel 175 mg/m^2, infusion, intravenously, once on Day 1 of 21-day cycle, followed by pevonedistat 20 mg/m^2, infusion, intravenously alone once on Days 3 and 5 in each 21-day cycle for up to 17 cycles or symptomatic deterioration or disease progression, treatment was discontinued for another reason, or until the study was stopped in Part B. Pevonedistat was administered after the paclitaxel and carboplatin chemotherapy. Participants who completed Part A and provided consent for Part B continued treatment in Part B.
Arm/Group | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg | Part B: Pevonedistat 25 mg/m^2 + Docetaxel 75 mg/m^2 | Part B: Pevonedistat 20 mg/m^2 + Carboplatin AUC5+ Paclitaxel 175 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/9 | 1/8
Serious Adverse Events (participants affected / at risk) | 3/20 | 3/9 | 4/8
Other Adverse Events (participants affected / at risk) | 11/20 | 9/9 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg (N=20) | Part B: Pevonedistat 25 mg/m^2 + Docetaxel 75 mg/m^2 (N=9) | Part B: Pevonedistat 20 mg/m^2 + Carboplatin AUC5+ Paclitaxel 175 mg/m^2 (N=8)
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Pevonedistat 50 mg/m^2 + Rifampin 600 mg (N=20) | Part B: Pevonedistat 25 mg/m^2 + Docetaxel 75 mg/m^2 (N=9) | Part B: Pevonedistat 20 mg/m^2 + Carboplatin AUC5+ Paclitaxel 175 mg/m^2 (N=8)
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2
Fatigue (General disorders) | 3 | 5 | 2
Oedema peripheral (General disorders) | 2 | 2 | 1
Pyrexia (General disorders) | 2 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1
Headache (Nervous system disorders) | 2 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 1
Medical device site oedema (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 4 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 4
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT03486314/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT03486314/SAP_001.pdf